CLINICAL TRIAL: NCT04883983
Title: Open Label Placebo to Manage Pain in Total Joint Arthroplasty: A Feasibility Study
Brief Title: OLP to Manage Pain in TJA: A Feasibility Study
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was never initiated.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tapan Shirish Mehta, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300006920; UAB (Other Grant/Funding Number: UAB)
Record Dates: First submitted 2021-04-08; First posted 2021-05-12 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Opioid Dependence; Opioid Abuse
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pain Medication as Standardly Prescribed (Active Comparator): Patients will receive pain medication as standardly prescribed. Refills at the 2 week followup will be provided as per the standard treatment protocol.
  Interventions: Drug: Patient medication as standardly prescribed
- Open Label Placebo (Experimental): Initial post-op pain medication will be prescribed. On 2 week followup, refill request will be filled with an open label placebo.
  Interventions: Drug: Open Label Placebo

INTERVENTIONS:
Drug: Open Label Placebo — Pain medication will be prescribed per standard treatment for initial prescription. Pain medication request at followup will be filled with open label placebo. Pain assessment surveys will be used at 2, 6, and 12 week followups.
  Arms: Open Label Placebo
Drug: Patient medication as standardly prescribed — Pain medication will be prescribed per standard treatment for initial prescription. On request for additional pain medication, pain medication will be prescribed as per the standard protocol. Pain assessment surveys will be used at 2, 6, and 12 week followups.
  Arms: Pain Medication as Standardly Prescribed

SUMMARY:
Persistent opioid abuse presents a common yet under-recognized problem given the decreasing rates of morbidity and mortality following common elective surgical procedures, like total joint arthroplasty (TJA). Each year around 33-70% of patients seeking surgical procedures in the U.S. transition to persistent opioid use following elective surgery (such as TJA), primarily prescribed for post-operative pain management. Further, these patients are more likely to demand greater doses and for longer duration post-surgery due to maladaptive neurologic changes occurring in key areas of the brain. The purpose of this study is to see if it is feasible to use OLP (open label placebo) for post-operative pain management in the post TJA setting. In addition the investigators will also collect pilot data to compare key outcome measures (patient reported physical function related to osteoarthritis of the hip and knee, pain score, and health-related quality of life will be assessed) between the placebo and the Treatment-As-Usual (TAU) group over a 90-day post-operative period.

DETAILED DESCRIPTION:
The investigators will enroll 24 adults that have undergone primary total joint arthroplasty and are requesting additional pain medication at 2 weeks. Once informed, consented and enrolled, participants will be assessed, randomized to either open-label placebo (OLP) or treatment-as-usual (TUA). Participants will be informed on why the OLP may manage the symptoms of postoperative pain and the benefits of OLP vs an Opioid. Patients randomized to OLP will be given placebo pills at their 2 week follow-up appointment (baseline) if additional pain medication is requested. Patients will be instructed to utilize placebo pill in the same manner as their previous medication. If interested, the participant will be consented in clinic and a consent signed in person. Pain control, joint function, and quality of life assessment scores will be conducted at 2, 6, and 12 week follow-up visits in clinic. After randomization, the placebo group will receive a scripted orientation that mimics a typical patient-provider interaction when prescribing a pain medication, including the rationale for effectiveness and the importance of taking the placebo pills as prescribed.

Open-label placebo adherence will be assessed using pill count. The investigators will ask all participants to maintain their current treatment regimens over the course of the study. After 12 weeks, all participants will complete final assessments. Participants in the OLP group will be monitored in clinic to allow for additional pain control if required.

Study outcomes will be measured using SF-36 quality of life score, Visual Analog Scale, Hip disability and Osteoarthritis Outcome Score, and Knee disability and Osteoarthritis Outcome Score. The investigators will also collect information about potential moderators that would include demographic data (e.g., age, years since diagnosis, treatments, gender), use of disease modifying therapies (oral versus infusion), types of medications, total number of medications, history of opioid abuse, history of opioid use, presence of a diagnosed cognitive or psychiatric disorder, mood disorder.

ANCOVA will be used to measure treatment effect with baseline measurement used as a covariate. Effect sizes and estimates of correlation between pre-post measures will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible to undergo the TJA surgical procedure

Exclusion Criteria:

* Participants who are not eligible to undergo the TJA surgical procedure i.e. (participants who are morbidly obese or with comorbidities that make them ineligible for the surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients with acceptable pain control as measured by Visual Analogue scale | 2 weeks (Baseline)
  VAS is a patient measured scale to evaluate pain, on a scale of 1-10 with 10 being the worst pain.
Percentage of Patients with acceptable pain control as measured by Visual Analogue scale | 6 weeks
  VAS is a patient measured scale to evaluate pain, on a scale of 1-10 with 10 being the worst pain.
Percentage of Patients with acceptable pain control as measured by Visual Analogue scale | 12 weeks
  VAS is a patient measured scale to evaluate pain, on a scale of 1-10 with 10 being the worst pain.
Percentage of Patients with acceptable quality of life as measured by Short Form Health Survey SF-36 | Week 2 (Baseline)
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Percentage of Patients with acceptable quality of life as measured by Short Form Health Survey SF-36 | Week 6
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Percentage of Patients with acceptable quality of life as measured by Short Form Health Survey SF-36 | Week 12
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Percentage of Patients with acceptable joint functionality as measured by knee disability and osteoarthritis outcome score (KOOS) | Baseline 2 weeks
  Knee disability and osteoarthritis outcome score (KOOS) is a patient measured score evaluating Knee function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by knee disability and osteoarthritis outcome score (KOOS) | 6 weeks
  Knee disability and osteoarthritis outcome score (KOOS) is a patient measured score evaluating Knee function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by knee disability and osteoarthritis outcome score (KOOS) | 12 weeks
  Knee disability and osteoarthritis outcome score (KOOS) is a patient measured score evaluating Knee function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by hip disability and osteoarthritis outcome score (HOOS). | Baseline 2 weeks
  Hip disability and osteoarthritis outcome score (HOOS) is a patient measured score evaluating Hip function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by hip disability and osteoarthritis outcome score (HOOS). | 6 weeks
  Hip disability and osteoarthritis outcome score (HOOS) is a patient measured score evaluating Hip function and creates a score out of 100, 100 indicating full functionality.
Percentage of Patients with acceptable joint functionality as measured by hip disability and osteoarthritis outcome score (HOOS). | 12 weeks
  Hip disability and osteoarthritis outcome score (HOOS) is a patient measured score evaluating Hip function and creates a score out of 100, 100 indicating full functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Naranje, Principal Investigator — University of Alabama at Birmingham; Tapan Mehta, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No